CLINICAL TRIAL: NCT07399340
Title: A Comparative Evaluation of the Role of Self-Adhesive Flowable Composite in Enhancing Sealant Retention Versus Conventional Pits and Fissure Sealant With and Without Fissurotomy in Permanent Molars: A Randomized Controlled Trial
Brief Title: A Comparative Evaluation of the Role of Self-Adhesive Flowable Composite in Enhancing Sealant Retention Versus Conventional Pits and Fissure Sealant With and Without Fissurotomy in Permanent Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Eman Mohamed Mostafa Ramadan, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CU-Pedo-2026
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pits and Fissure Sealants
Keywords: Self-adhering flowable composite; Conventional pits and fissure sealant; Helioseal-F; Vertise Flow; Fissurotomy; Permanent molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The blinding of the operator is not possible due to the nature of the materials used and fissurotomy preparation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self adhering flowable composite Vertise™ Flow with fissurotomy (Experimental): Vertise™ Flow (Kerr, Orange, CA, USA)
  Chemical composition:
  * Resin: GPDMA, HEMA, BisGMA, catalysts.
  * Fillers: Prepolymers, silanated Ba-glass, SiO2,YF3 (70 wt%). This SAFC uses the adhesive monomer glycerophosphate dimethacrylate GPDM, a phosphate functional group that creates a chemical bond with the calcium ions of the tooth. GPDM monomers ensure a tenacious bond to enamel, evidenced by the strength known to all generations of the OptiBond adhesive family.
  Interventions: Other: Self adhering flowable composite Vertise™ Flow (Kerr, Orange, CA, USA) with fissurotomy.
- Self adhering flowable composite Vertise™ Flow without fissurotomy (Experimental): Vertise™ Flow (Kerr, Orange, CA, USA)
  Chemical composition:
  * Resin: GPDMA, HEMA, BisGMA, catalysts.
  * Fillers: Prepolymers, silanated Ba-glass, SiO2,YF3 (70 wt%). This SAFC uses the adhesive monomer glycerophosphate dimethacrylate GPDM, a phosphate functional group that creates a chemical bond with the calcium ions of the tooth. GPDM monomers ensure a tenacious bond to enamel, evidenced by the strength known to all generations of the OptiBond adhesive family.
  Interventions: Other: Self adhering flowable composite Vertise™ Flow (Kerr, Orange, CA, USA) without fissurotomy.
- Conventional resin-based pits and fissure sealant Helioseal-F with fissurotomy. (Active Comparator): Resin-based pits and fissure sealant Helioseal-F 40% filler content, higher viscosity
  Sealant Matrix Composition:
  1. Bis-GMA
  2. UDMA
  3. TEGDMA Fillers: Fluorosilicate glass , highly dispersed silicon dioxide, pigments, initiators.
  Interventions: Other: Conventional resin-based pits and fissure sealant Helioseal-F with fissurotomy.
- Conventional resin-based pits and fissure sealant Helioseal-F without fissurotomy. (Active Comparator): Resin-based pits and fissure sealant Helioseal-F 40% filler content, higher viscosity
  Sealant Composition:
  1. Bis-GMA
  2. UDMA
  3. TEGDMA Fillers: Fluorosilicate glass , highly dispersed silicon dioxide, pigments, initiators.
  Interventions: Other: Conventional resin-based pits and fissure sealant Helioseal-F without fissurotomy.

INTERVENTIONS:
Other: Self adhering flowable composite Vertise™ Flow (Kerr, Orange, CA, USA) with fissurotomy. — 1. Pits and fissures will be prepared using a Micro STF fissurotomy bur (SS White Burs Inc., Lakewood, NJ, USA) on a high-speed hand piece, the bur will be moved along all the occlusal fissures with a gentle force applied. (Bagherian et al., 2013)
  2. Then washing and drying the tooth with compressed air.
  3. Then self-adhering flowable composite (Vertise Flow, Kerr, Orange, CA, USA) with an A2 shade will be applied on occlusal fissures in 0.5mm and brushed on preparation for 15-20sec using a micro-brush with moderate pressure. (Sabbagh et al., 2017; Sharma et al., 2018)
  4. Excess material around the margins will be removed.
  5. After ensuring that there are no bubbles, the sealant will be cured for 20 seconds by light cure. (Woodpecker RTA Mini S, China).
  6. If necessary, another layer will be applied and cured for 20 seconds.
  Arms: Self adhering flowable composite Vertise™ Flow with fissurotomy
Other: Self adhering flowable composite Vertise™ Flow (Kerr, Orange, CA, USA) without fissurotomy. — 1. Before applying Vertise Flow, surface pretreatment according to the manufacturers' recommendations for uncut enamel.(Kucukyilmaz and Savas, 2015) Using 37.5 % phosphoric acid gel Ivoclar Vivadent AG, Schaan, Liechtenstein) for 30-60 seconds according to the manufacturer's instructions, rinsed for 60 seconds and air-dried with oil- and water-free air spray using clean compressed air until observing the chalky white appearance.
  2. Then self-adhering flowable composite (Vertise Flow, Kerr, Orange, CA, USA) with an A2 shade will be applied in 0.5mm and brushed on fissures for 15-20sec using a micro-brush with moderate pressure.(Sabbagh et al., 2017; Sharma et al., 2018)
  3. Remove excess material around the margins.
  4. After ensuring that there are no bubbles, the sealant will be cured for 20 seconds by light cure. (Woodpecker RTA Mini S, China).
  5. If necessary, another layer will be applied and cured for 20 seconds.
  Arms: Self adhering flowable composite Vertise™ Flow without fissurotomy
Other: Conventional resin-based pits and fissure sealant Helioseal-F with fissurotomy. — 1. Pits and fissures will be prepared using a Micro STF fissurotomy bur (SS White Burs Inc., Lakewood, NJ, USA) on a high-speed hand piece, the bur will be moved along all the occlusal fissures with a gentle force applied. (Bagherian et al., 2013)
  2. Then the occlusal surface of the teeth will be dried and etched with 37% phosphoric acid (Ivoclar Vivadent AG, Schaan, Liechtenstein) for 15-30 seconds according to the manufacturer's instructions, rinsed for 30 seconds and air-dried with oil- and water-free air spray using clean compressed air until observing the chalky white appearance.
  3. Helioseal-F sealant (Ivoclar Vivadent AG, Schaan, Liechtenstein) will be applied and directed into the pits and fissures by a sterile explorer to check that there are no air bubbles and light cured for 40 seconds by light cure. (Woodpecker RTA Mini S, China).
  Arms: Conventional resin-based pits and fissure sealant Helioseal-F with fissurotomy.
Other: Conventional resin-based pits and fissure sealant Helioseal-F without fissurotomy. — 1. The occlusal surface of the teeth will be dried and etched with 37% phosphoric acid (Ivoclar Vivadent AG, Schaan, Liechtenstein) for 30-60 seconds according to the manufacturer's instructions, rinsed for 30 seconds and air-dried with oil- and water-free air spray using clean compressed air until observing the chalky white appearance.
  2. Helioseal-F sealant (Ivoclar Vivadent AG, Schaan, Liechtenstein) will be applied and directed into the pits and fissures by a sterile explorer to check that there are no air bubbles and light cured for 40 seconds by light cure. (Woodpecker RTA Mini S, China )
  Arms: Conventional resin-based pits and fissure sealant Helioseal-F without fissurotomy.

SUMMARY:
This RCT study aims to establish evidence-based decision comparing between self-adhering flowable composite Vertise™ Flow (Kerr, Orange, CA, USA) and conventional resin-based pits & fissure sealant Helioseal-F sealant (Ivoclar Vivadent AG, Schaan, Liechtenstein) with and without fissurotomy in sealant retention and prevention of occlusal pits and fissures caries in first permanent molars over a 12-month follow-up.

DETAILED DESCRIPTION:
This randomized controlled clinical trial aims to compare the retention and clinical performance of a self-adhering flowable composite and a conventional resin-based pit and fissure sealant, applied with and without fissurotomy, in newly erupted permanent first molars of children aged 6-8 years.

Occlusal pits and fissures are highly susceptible to dental caries in children, and long-term sealant effectiveness is strongly dependent on material retention and technique sensitivity. Self-adhering flowable composites offer simplified application with fewer clinical steps and may improve retention, especially in pediatric patients.

Eighty-eight children will be randomly allocated into four parallel groups (1:1:1:1): self-adhering flowable composite with fissurotomy, self-adhering flowable composite without fissurotomy, conventional resin-based sealant with fissurotomy, and conventional resin-based sealant without fissurotomy.

Sealant retention will be assessed as the primary outcome using Simonsen's criteria, while secondary outcomes include caries development, marginal discoloration, and marginal integrity evaluated using Ryge criteria.

Clinical evaluations will be performed at baseline, 3, 6, and 12 months.

The findings of this study aim to provide evidence-based guidance on the optimal material and technique for pit and fissure sealing in children, potentially improving sealant longevity, reducing occlusal caries incidence, and enhancing preventive pediatric dental care.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy children aged 6 to 8 years.
* Children with high caries risk
* Completely erupted lower first permanent molars with deep pits and fissures.
* Fissures either intact, sound or retentive which are stained, caries free or ICDAS 0-2.
* Availability for the duration of the study.
* Satisfactory dental care performed at home.

Exclusion Criteria:

* Children whose parents refuse to sign informed consent.
* Long-term medication affecting the salivary flow.
* Children enrolled for other studies or fluoridation program.
* Adverse reaction reported to any dental material.
* Uncooperative child.
* Bruxism or malocclusion.
* Children with developmental defects/ hypoplastic molars or caries affected teeth (ICDAS>2).
* Teeth with restoration and partially retained sealants.
* Children who cannot come for the follow-up.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Sealant retention | 3,6,12 months
  Simonsen's criteria Score 1: Complete retention Score 2: Partial loss Score 3: Complete loss

SECONDARY OUTCOMES:
Presence of Caries | 3,6,12 months
  Ryge criteria Alpha: Absence of caries Bravo: Prescence of caries
Marginal discoloration | 3,6,12 months
  Ryge criteria Alpha: No discoloration anywhere on the margin around the sealant. Bravo: Visible partial discoloration on the margin around sealant. Charlie: Visible discoloration on the margin around all sealant.
Marginal Integrity | 3,6,12 months
  Ryge criteria Alpha: Sealant had full adaptation to the adjacent tooth structure. Bravo: Evidence of gap detected by the tip of an explorer.

CONTACTS AND LOCATIONS:
Overall Officials: Adel ELbardissy, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, State/Province *, Egypt

IPD SHARING:
Plan to Share IPD: No